CLINICAL TRIAL: NCT00634959
Title: An Investigation Into The Effects Of Food And Dose Regimen On Viral Load Response In HIV Infected Patients On Short-Term Monotherapy With UK-427,857 (Maraviroc)
Brief Title: Effects Of Food And Dose Regimen On The Antiviral Effects Of Maraviroc (UK-427,857) In Patients With Human Immunodeficiency Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4001015
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: HIV
Keywords: HIV Infections; Treatment Naïve
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: Maraviroc (UK-427,857)
- 2 (Experimental)
  Interventions: Drug: Maraviroc (UK-427,857)
- 3 (Experimental)
  Interventions: Drug: Maraviroc (UK-427,857)
- 4 (Experimental)
  Interventions: Drug: Maraviroc (UK-427,857)
- 5 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Maraviroc (UK-427,857) — 150 mg oral tablet twice daily while fasted on Days 1-9 and on Day 10 (morning dose only)
  Other Names: Celsentri, Selzentry
  Arms: 1
Drug: Maraviroc (UK-427,857) — 100 mg oral tablet once daily while fasted on Days 1-10
  Other Names: Celsentri, Selzentry
  Arms: 2
Drug: Maraviroc (UK-427,857) — 300 mg oral tablet once daily while fasted on Days 1-10
  Other Names: Celsentri, Selzentry
  Arms: 3
Drug: Maraviroc (UK-427,857) — 150 mg oral tablet twice daily with food on Days 1-9 and on Day 10 (morning dose only)
  Other Names: Celsentri, Selzentry
  Arms: 4
Other: Placebo — Matching placebo oral tablet on Days 1-10 (fed and fasted)
  Arms: 5

SUMMARY:
To investigate the effects of food and dose regimen on the antiviral effects of Maraviroc (UK-427,857) in patients with human immunodeficiency virus (HIV)

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic HIV-1 infected male and female patients
* Weight between 50 and 100kg and within the permitted range for their height
* Patients with virus that targets CCR5 receptor

Exclusion Criteria:

* Patients with a CD4 count <250 cells/mm3 or HIV viral load <5000 copies/mL
* Patients whose HIV infection has been diagnosed less than 3 months prior to screening, or for who there is evidence of recent seroconversion
* Patients with acquired immunodeficiency syndrome (AIDS) or a previous AIDS diagnosis
* Patients who are taking or have taken antiretroviral drugs in the eight weeks prior to the study screening visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2003-07; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in viral load | Day 11
UK-427,857 pharmacokinetics | Days 1-11

SECONDARY OUTCOMES:
Physical examination | Days 1, 11, 40
12-lead ECG | Days 1-11 and Day 40
Relationship of change in viral load (baseline to Day 11) versus mean receptor saturation (Day 10) | Days 1-11
Time course of viral load from baseline to follow-up | Days 1-13 and Days 15, 19, 22, 25, 40
CCR5 receptor saturation | Days 1, 5, 10, 11, 13, 15, 19, 40
Adverse events | Days 1-40
Relationship of change in viral load (baseline to Day 11) versus baseline susceptibility (IC50 and IC90) | Days 1-11
Laboratory safety | Days 1, 3, 7, 11, 15, 40
Relationship of change in viral load (baseline to Day 11) versus average and trough plasma concentrations (Day 10) | Days 1-11
Supine/standing blood pressure and pulse rate | Days 1-11 and Day 40
Time to rebound of viral load | Days 1-13 and Days 15, 19, 22, 25, 40

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (2):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Boston, Massachusetts
- Germany (3):
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Hamburg
- Pfizer Investigational Site, London, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001015&StudyName=Effects%20Of%20Food%20And%20Dose%20Regimen%20On%20The%20Antiviral%20Effects%20Of%20Maraviroc%20%28UK-427%2C857%29%20In%20Patients%20With%20Human%20Immunodeficiency%20Virus